CLINICAL TRIAL: NCT05511350
Title: An Expanded Access Protocol for Subjects With Relapsed or Refractory Advanced Solid Tumors Receiving TJ210001
Brief Title: Expanded Access Protocol for Subjects With Relapsed or Refractory Advanced Solid Tumors Receiving TJ210001
Status: No longer available | Type: Expanded Access
Sponsor: I-Mab Biopharma US Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: TJ210001STM103
Record Dates: First submitted 2022-08-19; First posted 2022-08-23 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Solid Tumor Metastatic Cancer Advanced Cancer
Keywords: monoclonal antibody anti-C2aR

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: TJ210001

SUMMARY:
This EAP was designed to provide TJ210001 to the remaining subjects with relapsed or refractory solid tumors who were enrolled on the parent study, TJ210001STM101 (NCT04678921), and plan to continue with treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, of any race, age ≥ 18 years;
2. Participation in the parent TJ210001STM101 study and thought to have potential to derive clinical benefit from continued treatment in the opinion of the parent study investigator from uninterrupted dosing of TJ210001;
3. Willingness and ability to comply study treatment and standard of care testing and procedures;
4. Women of childbearing potential (WOCBP) must:

   1. Agree to use at least 2 effective contraceptive methods (1 highly effective method in combination with a barrier method; oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner), one of which must be barrier, from signing the ICF, throughout the study, and for up to 12 weeks following the last dose of TJ210001;
   2. Avoid conceiving for 12 weeks after the last dose of TJ210001;
   3. Avoid donation of ova until 12 weeks after the last dose of TJ210001;
   4. Agree to ongoing urine pregnancy testing, if clinically indicated, during the course of the study.
5. Males must agree to use a condom (a latex condom is recommended) during sexual contact with a pregnant female or a female of childbearing potential and will avoid donation of sperm or having a female partner conceive from the time of signing the ICF, while participating in the study, during dose interruptions, and for at least 12 weeks after the last dose of study treatment, even if he has undergone a successful vasectomy;
6. Patient or patient's health care proxy is able and willing to provide written informed consent and able to follow study instructions.

Exclusion Criteria:

* Any unresolved ongoing toxicity or clinical event that would make continued treatment with TJ210001 inappropriate; 2. Current treatment on another therapeutic clinical trial; 3. Currently pregnant; 4. Current evidence of any condition (including medical, psychiatric or substance abuse disorder), therapy, or laboratory abnormality that might interfere with the patient's participation or is not in the best interest of the patient to participate, in the opinion of the treating Investigator

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Laura Feller, NP, Principal Investigator — Horizon Oncology Center